CLINICAL TRIAL: NCT03653000
Title: Assessement of a Novel Approach to Ultrasound-guided Brachial Plexus Blockade, Located Between the Infraclavicular and the Axillary Site
Brief Title: Assessement of a Novel Approach to Ultrasound-guided Brachial Plexus Blockade
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, J P Lecoq, Medical Doctor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2018-07-27; First posted 2018-08-31 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Nerve Block
Keywords: Regional anesthesia; Ultrasound guided brachial plexus blockade; Local anesthetics : Ropivacaine
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Descriptive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing this new block (Experimental): Descriptive study about the effectiveness and the feasability of this new approach of te ultrasound guided brachial plexus blockade
  Interventions: Procedure: Ultrasound guided brachial plexus blockade; Drug: local anaesthetic injection

INTERVENTIONS:
Procedure: Ultrasound guided brachial plexus blockade — Ultrasound probe disposed on the shoulder, on the deltoid muscle. in plane puncture toward the brachial artery and injection of local anaesthetics around the brachial artery
Drug: local anaesthetic injection — Local anesthetic injection (ropivacaine) at this new site

SUMMARY:
Assessement of a new approach of an ultrasound guided brachial plexus blockade between the infraclavicular and axillary area.

DETAILED DESCRIPTION:
After an assessement of this new approach of ultrasounded-guided brachial plexus blockade in cadavers, the aim of this human study was to asssess the validity of this method in humans. The probe will be disposed on the shoulder, and the brachial plexus will be seeked below the deltoid, lateral to the major pectoralis muscle and in the vicinity of the brachial artery. At this area, an ultrasounded guided needle was inserted with an in-plane direction towards the brachial artery and local anesthetics was disposed all around the artery, without puncturing the differents nerves. Regional blockade will be evaluated by measuring onset and duation time for sensitive and motor blockade, effectiveness of this blockade, patient's confort during the procedure, ease of the procedure for practitionner, quality of ultrasound image's interpretation before and after injection.

ELIGIBILITY:
Inclusion Criteria:

* Arm surgery performed under axillary blockade

Exclusion Criteria:

* Local anesthetics allergy
* Coagulation disorder
* History of chronic pain
* Drug or alcohol abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of block realisation assessed by number of abandonned block | Immediately after procedure
  Difficulty in the block realisation (block abandonned before or during realisation)
Efficience of the block assessed by number of block sufficient for surgery | Immediately after procedure
  Is the block enough for surgery or must be completed
Comfort during block realization assessed by Numeric Rating Scale (NRS - 0 = No pain, 10 = worse pain) | Immediately after procedure
  Evaluation of comfort during block realization
Evaluation of motor block for the median nerve at 5 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 5 minutes post injection
  Evaluation of motor block for the median nerve
Evaluation of motor block for the median nerve at 10 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 10 minutes post injection
  Evaluation of motor block for the median nerve
Evaluation of motor block for the median nerve at 15 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 15 minutes post injection
  Evaluation of motor block for the median nerve
Evaluation of motor block for the median nerve at 20 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 20 minutes post injection
  Evaluation of motor block for the median nerve
Evaluation of motor block for the ulnar nerve at 5 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 5 minutes post injection
  Evaluation of motor block for the ulnar nerve
Evaluation of motor block for the ulnar nerve at 10 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 10 minutes post injection
  Evaluation of motor block for the ulnar nerve
Evaluation of motor block for the ulnar nerve at 15 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 15 minutes post injection
  Evaluation of motor block for the ulnar nerve
Evaluation of motor block for the ulnar nerve at 20 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 20 minutes post injection
  Evaluation of motor block for the ulnar nerve
Evaluation of motor block for the radial nerve at 5 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 5 minutes post injection
  Evaluation of motor block for the radial nerve
Evaluation of motor block for the radial nerve at 10 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 10 minutes post injection
  Evaluation of motor block for the radial nerve
Evaluation of motor block for the radial nerve at 15 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 15 minutes post injection
  Evaluation of motor block for the radial nerve
Evaluation of motor block for the radial nerve at 20 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 20 minutes post injection
  Evaluation of motor block for the radial nerve
Evaluation of motor block for the musculocutaneous nerve at 5 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 5 minutes post injection
  Evaluation of motor block for the musculocutaneous nerve
Evaluation of motor block for the musculocutaneous nerve at 10 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 10 minutes post injection
  Evaluation of motor block for the musculocutaneous nerve
Evaluation of motor block for the musculocutaneous nerve at 15 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 15 minutes post injection
  Evaluation of motor block for the musculocutaneous nerve
Evaluation of motor block for the musculocutaneous nerve at 20 minutes post injection assessed by a scale of motor function (0 = Complete paresis, 1 = Partial paresis, 2 = Normal motion) | 20 minutes post injection
  Evaluation of motor block for the musculocutaneous nerve
Evaluation of sensitive block for the median nerve at 5 minutes post injection assessed by a scale of sensitive function (0 = No sensibility, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 5 minutes post injection
  Evaluation of sensitive block for the median nerve at 5 minutes post injection
Evaluation of sensitive block for the median nerve at 10 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 10 minutes post injection
  Evaluation of sensitive block for the median nerve at 10 minutes post injection
Evaluation of sensitive block for the median nerve at 15 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 15 minutes post injection
  Evaluation of sensitive block for the median nerve at 15 minutes post injection
Evaluation of sensitive block for the median nerve at 20 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 20 minutes post injection
  Evaluation of sensitive block for the median nerve at 20 minutes post injection
Evaluation of sensitive block for the ulnar nerve at 5 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 5 minutes post injection
  Evaluation of sensitive block for the ulnar nerve at 5 minutes post injection
Evaluation of sensitive block for the ulnar nerve at 10 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 10 minutes post injection
  Evaluation of sensitive block for the ulnar nerve at 10 minutes post injection
Evaluation of sensitive block for the ulnar nerve at 15 minutes post injection (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 15 minutes post injection
  Evaluation of sensitive block for the ulnar nerve at 15 minutes post injection
Evaluation of sensitive block for the ulnar nerve at 20 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 20 minutes post injection
  Evaluation of sensitive block for the ulnar nerve at 20 minutes post injection
Evaluation of sensitive block for the radial nerve at 5 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 5 minutes post injection
  Evaluation of sensitive block for the radial nerve at 5 minutes post injection
Evaluation of sensitive block for the ulnar nerve at 15 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 15 minutes post injection
  Evaluation of sensitive block for the ulnar nerve at 15 minutes post injection
Evaluation of sensitive block for the musculocutaneous nerve at 5 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 5 minutes post injection
  valuation of sensitive block for the musculocutaneous nerve at 5 minutes post injection
Evaluation of sensitive block for the musculocutaneous nerve at 10 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 10 minutes post injection
  Evaluation of sensitive block for the musculocutaneous nerve at 10 minutes post injection
Evaluation of sensitive block for the musculocutaneous nerve at 15 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 15 minutes post injection
  Evaluation of sensitive block for the musculocutaneous nerve at 15 minutes post injection
Evaluation of sensitive block for the musculocutaneous nerve at 20 minutes post injection assessed by a scale of sensitive function (0 = No sensibilityto cold, 1 = partial insensibility to cold, 2 = Normal sensation to cold) | 20 minutes post injection
  Evaluation of sensitive block for the musculocutaneous nerve at 20 minutes post injection

SECONDARY OUTCOMES:
Demographic data AGE | At the time of the procedure
  Age of the patient
Demographic data WEIGHT | At the time of the procedure
  Weight of the patient
Demographic data HEIGHT | At the time of the procedure
  Height of the patient
Type of surgery | At the time of the procedure
  hand surgery on bone/tendon/ligament/skin/nerve
Tourniquet | At the time of the procedure
  Time of tourniquet during surgery
Type of hospitalization | At the time of the procedure
  One or more day hospitalization
Local anesthetics used | At the time of the procedure
  Amount of local anesthetics used
Operator impression | At the time of the procedure
  Impression of the difficulty for the operator to perform the block
Incident during block performance | At the time of the procedure
  Incidence during block performance
Duration of block performance | At the time of the procedure
  Time of block performance
Duration of motor block | from 0 to day 1
  duration of motor block
Duration of sensitive block | from 0 to day 1
  duration of sensitive block
Block injury | From day 0 to day 7
  Neuropathy or other secondary effect post block during 7 days
Comparative image axillary and novel point of puncture | During the procedure
  Number of halo separating artery from different nerves at this novel level and at the axillary level

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Guntz Emmanuel, Braine-l'Alleud, Brabant Wallon
  - Lecoq Jean-Pierre, Liège, Liege

IPD SHARING:
Plan to Share IPD: No
No sharing data